CLINICAL TRIAL: NCT06191796
Title: A Phase 1b/2 Dose-finding and Expansion Study Evaluating the Safety and Efficacy of Zanzalintinib (XL092) Combined With Either AB521 or AB521 Plus Nivolumab in Subjects With Advanced Clear Cell Renal Cell Carcinoma or Other Advanced Solid Tumors.
Brief Title: Study of Zanzalintinib (XL092) + AB521 and Zanzalintinib + AB521 + Nivolumab in Participants With Advanced Clear Cell Renal Cell Carcinoma (ccRCC) or Other Advanced Solid Tumors (STELLAR-009)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study was terminated prior to starting the Phase 2 portion due to a business decision.
Sponsor: Exelixis (Industry)
Collaborators: Arcus Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XL092-009
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Advanced Clear Cell Renal Cell Carcinoma or Other Advanced Solid Tumors
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-finding Cohort A: Zanzalintinib + AB521 (Experimental): Participants with solid tumors will receive zanzalintinib + AB521
  Interventions: Drug: zanzalintinib; Drug: AB521
- Dose-finding Cohort B: zanzalintinib + AB521 + nivolumab (Experimental): Participants with ccRCC will receive zanzalintinib + AB521 + nivolumab
  Interventions: Drug: zanzalintinib; Drug: AB521; Biological: Nivolumab
- Expansion Cohort 1: Zanzalintinib + AB521 (Experimental): Participants with ccRCC will receive zanzalintinib + AB521
  Interventions: Drug: zanzalintinib; Drug: AB521
- Expansion Cohort 2: zanzalintinib + AB521 + nivolumab (Experimental): Participants with ccRCC will receive zanzalintinib + AB521 + nivolumab
  Interventions: Drug: zanzalintinib; Drug: AB521; Biological: Nivolumab

INTERVENTIONS:
Drug: zanzalintinib — Specified doses on specified days
  Other Names: XL092
Drug: AB521 — Specified doses on specified days
Biological: Nivolumab — Specified doses on specified days
  Other Names: OPDIVO®
  Arms: Dose-finding Cohort B: zanzalintinib + AB521 + nivolumab; Expansion Cohort 2: zanzalintinib + AB521 + nivolumab

SUMMARY:
The goal of this clinical trial is to learn about the safety and preliminary antitumor activity of zanzalintinib in combination with AB521 (doublet) and in combination with AB521 plus nivolumab (triplet) in participants with advanced ccRCC or other advanced solid tumors. The main questions it aims to answer are:

* The recommended doses (RDs)
* The safety and tolerability
* The PK and the preliminary efficacy

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with a).unresectable advanced or metastatic solid tumor; b). unresectable advanced or metastatic clear cell renal cell carcinoma and no prior anticancer therapy; or c). unresectable advanced or metastatic clear cell renal cell carcinoma and has received at least one prior anticancer therapy.
2. Measurable disease according to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1; Eisenhauer et al, 2009) as determined by the Investigator.
3. For all participants, archival tumor tissue material should be obtained; if archival tissue is not available or is older than 2 years, then a fresh biopsy should be obtained, if medically feasible. Specific requirements for tumor tissue samples will be described in the Laboratory Manual.
4. Recovery to baseline or ≤ Grade 1 per Common Terminology Criteria for Adverse Events (CTCAE) v5 from AE(s) related to any prior treatments unless AE(s) are deemed clinically nonsignificant by the Investigator and/or stable on supportive therapy.
5. Karnofsky Performance Status (KPS) ≥70%.
6. Screening ambulatory oxygen saturation (SpO2) ≥92%.
7. Screening left ventricular ejection fraction (LVEF) above the institutional lower limit of normal.

Key Exclusion Criteria:

1. Participants who have been previously treated with a HIF-2α targeted therapy and/or zanzalintinib.
2. Radiation therapy for bone metastases within 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Participants with clinically-relevant ongoing complications from prior radiation therapy are not eligible.
3. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery (including radiosurgery) and stable for at least 4 weeks before first dose of study treatment.
4. Concomitant anticoagulation with oral anticoagulants except for a). prophylactic use of low-dose aspirin for cardioprotection or low dose low molecular weight heparins (LMWH) or b). therapeutic doses of LMWH or specified direct factor Xa inhibitors.
5. Administration of a live, attenuated vaccine within 30 days prior to enrollment.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-01-25 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Dose-finding Stage: Number of participants with dose-limiting toxicities (DLTs) | Up to 24 months
Expansion Stage: Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the Investigator | Up to 24 months

SECONDARY OUTCOMES:
Dose-finding Stage: Number of participants with adverse events (AEs), including serious adverse events (SAEs) and immune-mediated adverse events (imAEs) | Up to 24 months
Dose-finding Stage: Concentration of study treatments (zanzalintinib and AB521) in plasma at specified time points | Up to 24 months
Dose-finding Stage: Objective response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 as assessed by the Investigator | Up to 24 months
Expansion Stage: Number of participants with adverse events (AEs), including serious adverse events (SAEs), and immune-mediated adverse events (imAEs) | Up to 24 months
Expansion Stage: Duration of response (DOR) per RECIST 1.1 as assessed by the Investigator | Up to 24 months
Expansion Stage: Progression-free survival (PFS) per RECIST 1.1 as assessed by the Investigator | Up to 24 months
Expansion Stage: Overall survival (OS) | Up to 24 months
Expansion Stage: Concentration of study treatments (zanzalintinib and AB521) in plasma at specified time points | Up to 24 months

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Exelixis Site #8, Los Angeles, California
  - Exelixis Site #9, Miami, Florida
  - Exelixis Clinical Site #1, Orlando, Florida
  - Exelixis Site #11, Tampa, Florida
  - Exelixis Site #6, Scarborough, Maine
  - Exelixis Site #5, St Louis, Missouri
  - Exelixis Clinical Site #3, New Hyde Park, New York
  - Exelixis Site #14, New York, New York
  - Exelixis Site #13, Shirley, New York
  - Exelixis Site #15, The Bronx, New York
  - Exelixis Clinical Site #2, Nashville, Tennessee
  - Exelixis Clinical Site #16, Salt Lake City, Utah
  - Exelixis Site #4, Spokane, Washington
  - Exelixis Site #12, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No